CLINICAL TRIAL: NCT04262401
Title: Habit Design: Testing a Novel Behavioral Approach to Corporate Wellness in the Context of Metabolic Syndrome
Brief Title: Promoting Healthy Habits in Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Habit Design (Industry)
Collaborators: University of Washington (Other); TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R44HL142328 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard health coaching (Active Comparator): Standard health coaching to increase health behaviors
  Interventions: Behavioral: Standard health coaching
- Habit-focused health coaching (Experimental): Health coaching enhanced with a focus on habit formation using a mobile application called Habit Design
  Interventions: Behavioral: Habit-focused health coaching

INTERVENTIONS:
Behavioral: Standard health coaching — 12 weekly sessions of standard health coaching followed by 4 monthly sessions
  Arms: Standard health coaching
Behavioral: Habit-focused health coaching — 12 weekly sessions of standard health coaching followed by 4 monthly sessions
  Arms: Habit-focused health coaching

SUMMARY:
A randomized controlled trial will be conducted to evaluate the effectiveness of the Habit Design (HD) approach in a corporate health context over the course of one year in subjects with metabolic syndrome. All subjects will be coached to increase physical activity. Additionally, subjects will choose and be coached to achieve a goal of either increasing fruit and vegetable intake or substituting water for sugar-sweetened beverages. Subjects will be randomly assigned to receive either standard coaching (control condition) or HD-enhanced coaching (experimental condition).

DETAILED DESCRIPTION:
To evaluate the effectiveness of the Habit Design approach, the investigators will conduct a randomized controlled trial with 424 corporate health program participants over the course of one year. Study subjects will be employees of TriHealth or their spouses who have completed a health screening as part of their corporate wellness program and identified as having metabolic syndrome. All subjects will be coached to increase physical activity, which will be monitored with a Fitbit and Fitabase software. Additionally, prior to randomization, subjects will choose a goal of increasing fruit and vegetable intake or substituting water for sugar-sweetened beverages. Subjects will be randomly assigned to receive either standard coaching (control condition) or HD-enhanced coaching (experimental condition). Conditions will be stratified/balanced by choice of goal and gender using urn randomization. In both conditions coaching will be manualized, monitored for fidelity, and delivered via telephone in 12 weekly active coaching sessions followed by 4 monthly maintenance coaching sessions. Coaching sessions will last 15-30 minutes. The primary outcome will be average daily step count measured with Fitbit over the course of at least one week at baseline, 16 weeks, 32 weeks, and 48 weeks. The secondary outcomes will be indices of fruit/vegetable intake or water intake, according to the participant's choice. Tertiary outcomes will consist of fasting blood glucose, triglycerides, high density lipoprotein, blood pressure, waist circumference, and body mass index, measured at each time point. Additionally, self-reported physical activity; junk food, and sugar-sweetened beverage consumption; automaticity of exercise and fruit, vegetable, and water consumption; self-efficacy and social support for target behaviors; and health-related quality of life will be assessed over time. Ratings of usability and satisfaction and app usage metrics will also be examined. Analyses will be intent-to-treat and assume 15% loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Participant in TriHealth's Corporate Wellness Program completing voluntary Personal Health Assessment, including screening for metabolic syndrome.
2. Meet at least 3/5 criteria for metabolic syndrome:

   * elevated triglycerides (≥150 mg/dL),
   * insufficient high-density lipoprotein cholesterol (<40 mg/dL in males and <50 mg/dL in females)
   * elevated blood pressure (systolic ≥130 and/or diastolic ≥85 mm Hg)
   * elevated fasting blood glucose (≥100 mg/dl)
   * above-threshold waist circumference (≥102 cm in males and ≥80 cm in females)
3. Interested in increasing physical activity and fruit/vegetable or water intake
4. Own a compatible smartphone (iOS or Android) and willing/able to use it for the study

Exclusion Criteria:

* Have medical or other contraindications to increasing physical activity or fruit/vegetable/water intake

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 424 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline average daily step count at 16 weeks | 16 weeks
  Fitbit data will be monitored using the Fitabase platform.
Change from baseline average daily step count at 32 weeks | 32 weeks
  Fitbit data will be monitored using the Fitabase platform.
Change from baseline average daily step count at 48 weeks | 48 weeks
  Fitbit data will be monitored using the Fitabase platform.

SECONDARY OUTCOMES:
Change in frequency consuming fruits and vegetables in the past 4 months at 16 weeks | 16 weeks
  Self-reported food frequency data derived from the Diet History Questionnaire-III. Fifteen items for fruits and fifteen items for vegetables will be rated on a scale from 0-9 and a sum of the item scores will be computed. Minimum: 0, Maximum: 270. Higher numbers are better.
Change in frequency consuming fruits and vegetables in the past 4 months at 32 weeks | 32 weeks
  Self-reported food frequency data derived from the Diet History Questionnaire-III. Fifteen items for fruits and fifteen items for vegetables will be rated on a scale from 0-9 and a sum of the item scores will be computed. Minimum: 0, Maximum: 270. Higher numbers are better.
Change in frequency consuming fruits and vegetables in the past 4 months at 48 weeks | 48 weeks
  Self-reported food frequency data derived from the Diet History Questionnaire-III. Fifteen items for fruits and fifteen items for vegetables will be rated on a scale from 0-9 and a sum of the item scores will be computed. Minimum: 0, Maximum: 270. Higher numbers are better.
Change in frequency consuming water in the past 4 months at 16 weeks | 16 weeks
  Self-reported food frequency data derived from the Diet History Questionnaire-III. Two items for water will be rated on a scale from 0-9 and a sum of the item scores will be computed. Minimum: 0, Maximum: 18. Higher numbers are better.
Change in frequency consuming water in the past 4 months at 32 weeks | 32 weeks
  Self-reported food frequency data derived from the Diet History Questionnaire-III. Two items for water will be rated on a scale from 0-9 and a sum of the item scores will be computed. Minimum: 0, Maximum: 18. Higher numbers are better.
Change in frequency consuming water in the past 4 months at 48 weeks | 48 weeks
  Self-reported food frequency data derived from the Diet History Questionnaire-III. Two items for water will be rated on a scale from 0-9 and a sum of the item scores will be computed. Minimum: 0, Maximum: 18. Higher numbers are better.
Change in baseline triglycerides at 16 weeks | 16 weeks
  Triglycerides will be measured using standard laboratory procedures.
Change in baseline triglycerides at 32 weeks | 32 weeks
  Triglycerides will be measured using standard laboratory procedures.
Change in baseline triglycerides at 48 weeks | 48 weeks
  Triglycerides will be measured using standard laboratory procedures.
Change in baseline fasting blood glucose at 16 weeks | 16 weeks
  Fasting blood glucose will be measured using standard laboratory procedures.
Change in baseline fasting blood glucose at 32 weeks | 32 weeks
  Fasting blood glucose will be measured using standard laboratory procedures.
Change in baseline fasting blood glucose at 48 weeks | 48 weeks
  Fasting blood glucose will be measured using standard laboratory procedures.
Change in baseline blood pressure at 16 weeks | 16 weeks
  Systolic and diastolic blood pressure will be measured using standard procedures.
Change in baseline blood pressure at 32 weeks | 32 weeks
  Systolic and diastolic blood pressure will be measured using standard procedures.
Change in baseline blood pressure at 48 weeks | 48 weeks
  Systolic and diastolic blood pressure will be measured using standard procedures.
Change in baseline waist circumference at 16 weeks | 16 weeks
  Waist circumference will be measured using standard procedures.
Change in baseline waist circumference at 32 weeks | 32 weeks
  Waist circumference will be measured using standard procedures.
Change in baseline waist circumference at 48 weeks | 48 weeks
  Waist circumference will be measured using standard procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kim, MBA, Principal Investigator — Habit Design; Susan Stoner, PhD, Principal Investigator — University of Washington; Scott Woods, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No